CLINICAL TRIAL: NCT06174064
Title: Broadband Light for the Treatment of Dry Eye Disease and Meibomian Gland Dysfunction
Brief Title: BroadBand Light for the Treatment of Dry Eye Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern California (Other)
Collaborators: Ophthalmic Surgeons & Consultants of Ohio, Inc. (Other)
Responsible Party: Principal Investigator, Sandy Zhang-Nunes, Director of Oculoplastics, USC Roski Eye Institute, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USCBBLDRYEYE
Record Dates: First submitted 2018-02-04; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye Syndromes; Meibomian Gland Dysfunction
Keywords: Dry eye; Blepharitis; Meibomian gland dysfunction; intense pulsed light
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction; Blepharitis | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to three arms: protocol 1, 2, and sham
Who Masked: Participant, Investigator
Masking Description: Patients will be randomized to protocol 1, 2, or sham but will not be aware of their assignment; investigators grading dry eye at baseline and after treatment will not be aware of which protocol the patients underwent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Protocol 1--420 and 560nm wavelengths (Active Comparator): Broadband light treatment Patients will be treated with BBL with 420nm wavelength filter followed by 560nm wavelength filter to malar and periorbital areas once monthly for 3 months. Dry eye evaluation consisting of clinical testing as well as quality of life questionnaires will be performed at baseline and after the last BBL treatment.
  Interventions: Device: Broadband Light treatment
- Protocol 2--560nm wavelength (Active Comparator): Broadband Light treatment Patients will be treated with BBL with 560nm wavelength filter to malar and periorbital areas once monthly for 3 months. Dry eye evaluation consisting of clinical testing as well as quality of life questionnaires will be performed at baseline and after the last BBL treatment.
  Interventions: Device: Broadband Light treatment
- Sham (Sham Comparator): Sham Broadband Light Treatment Patients will undergo the same preparation and procedure as for BBL treatment but the light source will be occluded. Patients will be treated with sham to malar and periorbital areas once monthly for 3 months. Dry eye evaluation consisting of clinical testing as well as quality of life questionnaires will be performed at baseline and after the last sham treatment.
  Interventions: Device: Sham broadband light treatment

INTERVENTIONS:
Device: Broadband Light treatment — While shielding the eyes, multiple passes of broadband light will be applied to the upper cheeks and eyelids after applying topical lidocaine.
  Other Names: Intense Pulsed Light
  Arms: Protocol 1--420 and 560nm wavelengths; Protocol 2--560nm wavelength
Device: Sham broadband light treatment — The light will be occluded on the usual BBL device so that no treatment is delivered but the preparation and procedure will otherwise be the same.
  Arms: Sham

SUMMARY:
The investigators will be evaluating the use of broadband light in Dry Eye and Meibomian Gland Dysfunction.

DETAILED DESCRIPTION:
Broadband light (BBL) is a widely used treatment for improvement of inflammatory dermatologic conditions such as acne and rosacea, and may have similar therapeutic benefits on the treatment of dry eye disease by targeting inflammation of the eyelids. The investigators propose a prospective study to determine the safety and efficacy of BBL treatment on patients with dry eye disease and meibomian gland dysfunction. Each participant will have three treatments of BBL at monthly intervals to the cheek and periorbital area with subsequent follow up. Measured endpoints will include signs and symptoms of dry eye control including full ophthalmic exam, dry eye diagnostic testing, photographs, and standardized questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I-V
* Must be diagnosed with Dry eye disease (DED) and meibomian gland dysfunction (MGD)
* Persistent dry eye signs and or symptoms after at least one prior DED treatment modality

Exclusion Criteria:

* Prior Intense pulsed light treatment for DED within the past six months
* Prior Meibomian gland treatment with a device for DED within the past three months
* History of trauma-induced ocular surface disease (thermal burns, chemical burns)
* Subject is pregnant
* History of seizures
* Having significant unprotected sun exposure within the treatment area
* Use of Accutane within the last six months
* Use of doxycycline in the last 1 month
* Allergy to proparacaine or lidocaine
* Having active herpes simplex virus infection within the treatment area
* Laser eye surgery (LASIK) within the past twelve months
* History of abnormal response to sunlight
* Having an active medical condition that may affect normal healing
* Having active infections or compromised immune system
* History of basal cell carcinoma in the treatment area within the past twelve months
* History of keloid scar formation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in dry eye score | 1 month after last BBL treatment (4 month time-point)
  Change in SPEED dry eye disease questionnaire score from baseline to 1 month post-treatment

SECONDARY OUTCOMES:
Ocular surface/eyelid microbiome data | 1 month after last BBL treatment
  genomic analysis of ocular surface flora at baseline compared to 1 month post-treatment
Clinical evaluation of dry eye-- Change in fluorescein staining grade | 1 month after last BBL treatment
  Change in Fluorescein staining graded with Oxford scale score from baseline to 1 month post-treatment
Clinical evaluation of dry eye--Change in tear osmolarity | 1 month after last BBL treatment
  Change in tear osmolarity (in milliosm/L) from baseline to 1 month post-treatment
Clinical evaluation of dry eye--Change in Matrix metalloproteinase-9 (MMP-9) presence in significant concentration | 1 month after last BBL treatment
  Change in MMP-9 testing (test is "positive" for MMP-9 level above 40ng/mL, and "negative" if below that threshold) from baseline to 1 month post-treatment
Clinical evaluation of dry eye--Change in tear breakup time | 1 month after last BBL treatment
  Change in tear break up time (in seconds) from baseline to 1 month post-treatment
Clinical evaluation of dry eye--Change in basal tear production | 1 month after last BBL treatment
  Change in basal tear production (in millimeters using standardized filter paper) from baseline to 1 month post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Zhang-Nunes, MD, Principal Investigator — USC Roski Eye Institute

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT06174064/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT06174064/SAP_001.pdf